CLINICAL TRIAL: NCT06569849
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Arm Clinical Trial of De-Stress and Focus Capsule in the Management of Stress, Mental Alertness, Fatigue, and Anxiety
Brief Title: A Clinical Trial of De-stress and Focus Capsule in the Management of Stress.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herbolab India Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MHC/CT/24-25/017; CTRI/2024/07/071243 (Registry Identifier: Clinical trials registry of India)
Record Dates: First submitted 2024-08-10; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Anxiety; Stress; Stuporous
Keywords: stress; Mental alertness; Fatigue; Anxiety
MeSH Terms: conditions — Anxiety Disorders; Stupor; Fatigue

STUDY DESIGN:
Intervention Model Description: Randomized, Double blind, Parallel Group, Placebo Controlled Trial
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- De-Stress and Focus capsule- U001 (Experimental)
  Interventions: Other: De-Stress and Focus capsule- U001
- De-Stress and Focus capsule - I001 (Experimental)
  Interventions: Other: De-Stress and Focus capsule - I001
- Placebo capsules 001 (Placebo Comparator)
  Interventions: Other: Placebo capsules 001

INTERVENTIONS:
Other: De-Stress and Focus capsule- U001 — Two capsules in sequence daily after meal for 60 days.
  Arms: De-Stress and Focus capsule- U001
Other: De-Stress and Focus capsule - I001 — Two capsules in sequence daily after meal for 60 days.
  Arms: De-Stress and Focus capsule - I001
Other: Placebo capsules 001 — Two capsules in sequence daily after meal for 60 days.
  Arms: Placebo capsules 001

SUMMARY:
The current study focuses in clinical validation of the efficacy of nutraceutical product in the management of mental focus and cognition. The benefits of these nutraceuticals extend beyond mere cognitive enhancement. Improved mental focus can lead to increased productivity and efficiency in both personal and professional settings. Individuals who struggle with attention deficits or cognitive fog may find that these supplements help them maintain a sharper and more consistent level of mental clarity. This can translate to better performance at work, as well as improved ability to manage daily tasks and responsibilities.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-arm clinical trial of De-Stress and Focus Capsule in the Management of Stress, Mental Alertness, Fatigue, and Anxiety

In this study, more than 60 participants will be enrolled and randomized to either one of the following groups: Group A: De-Stress and Focus Capsules-U001, Group B: De-Stress and Focus Capsules-I001, Group C: Placebo Capsules 001 in 1:1:1 ratio (20 patients in each group). The study duration is 60 days. The efficacy of the investigational products will be compared between the groups.

Concomitant diseases/medication assessment will be performed on screening.

Assessment of perceived stress scale (PSS) score, Montreal Cognitive Assessment (MoCA) scale score, Rey Complex Figure Test (RCFT), Trail Making Test (TMT) score, digit span memory test - forward and backward for attention and working memory assessment (most extended sequence), fatigue severity scale (FSS) score, mental chatter 5-point scale, Epworth Sleepiness Scale for daytime sleepiness, energy levels by using energy audit diary and adult ADHD Self-Report Scale (ASRS) score will be done at screening, day 30 and day 60.

Assessment of serum cortisol levels will be done at screening, day 15 and day 60.

Assessment of COPE Questionnaire (a. Positive Subscale b. Denial Subscale) score, STAI (State-Trait Anxiety Inventory) score, and Profile of Mood State (POMS) questionnaire score (a. Total Mood Disturbance b. Depression) will be done at screening and day 60.

Assessment of alertness, orientation, executive control functioning, and executive/arousal vigilance will be assessed using ANTI-Vea-UGR computerized test will be done at 0 hr, 1hr, 4 hr, and 8 hr after dosing on day 1, and day 60 (5 participants from each group i.e, total 15 participants).

Changes in vital sign parameters will be assessed from screening to the end of the study (Day 60). Assessment of changes in complete blood count, liver function test, and kidney function test will be done at screening and end of the study (Day 60). Safety of the investigational treatment in terms of adverse events (AEs), and serious adverse events (SAEs) from screening to end of the study ( Day 60). Treatment compliance and tolerability will be assessed from baseline to the end of the study (Day 60).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged 18-50 years both inclusive
2. Suffering from self-reported mild to moderate stress on the PSS scale score less than or equal to 26
3. Scoring 18-26 on the Montreal Cognitive Assessment MoCA
4. No or minimal impairment in activities of daily living: scoring less than 9 on the Functional Activities Questionnaire FAQ
5. Participants willing to participate in clinical trials and who have read understood and signed the informed consent form
6. No severe anxiety and depression on GAD and PHQ-9 scales
7. Able to complete the cognitive assessment tests

Exclusion Criteria:

1. Inability to perform any of the assessments required for endpoint analysis
2. Shows signs of Dementia, such as caused by Alzheimer's Disease, acquired immunodeficiency syndrome AIDS, Creutzfeldt-Jakob disease, Lewy Bodies dementia LBD, Cerebrovascular dementia CVD, Progressive Supranuclear Palsy PSP, multiple cerebral infarctions, or normal pressure hydrocephalus NPH, cardiac disease or endocrine disease
3. Have any other neurodegenerative diseases
4. History of a seizure disorder
5. Known hypersensitivity to investigational products
6. Participants with a history of malignancy diagnosed within the past 5 years or currently diagnosed with malignancy
7. Sitting or resting systolic blood pressure of more than 180 mm Hg or diastolic blood pressure of more than 110 mm Hg at Screening.
8. Participants with a history of substance abuse, drugs, heavy use of alcohol, and/or smoking within the last 5 years
9. Participants currently using medications and or supplements that could have cognitive or mood effects including but not limited to nutraceutical, allopathic, ayurvedic herbal extract or supplement
10. Pregnant or lactating women, as well as women of childbearing potential who are not using contraception or intending to conceive during the study
11. Serious illness or any other condition that, in the opinion of the investigator may compromise the safety or compliance of the patient or preclude the successful completion of the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-05 (Estimated); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale | Screening Baseline day 15 day 30 day 60
  The PSS-10 is widely used for measuring psychological distress. It contains 10 questions on a five-point scale from 0 to 4. The higher the score, the greater the feeling of stress. PSS-10 Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Montreal Cognitive Assessment (MoCA) | Screening, baseline, day 15, day 30, day 60
  Montreal Cognitive Assessment (MoCA) MoCA was a questionnaire performed preoperative then post-operative. The MoCA used in this study was developed by Professor Nasreddine in 2004 and is used for the rapid screening assessment of mild cognitive impairment. The cognitive areas assessed by MoCA included attention and concentration, executive function, memory, language, visual structure skills, abstract thinking, calculation and orientation. The scale had a total score of 30 points. ≥26 points were considered as having no cognitive impairment .
Rey Complex Figure Test (RCFT) | Screening, baseline, day 15, day 30, day 60
  The RCFT 'copy' is a validated, instrument assessing visuo-constructive abilities. The RCFT 'copy' requires the subject to observe and replicate an image. The score is scored as 0, 0.5, 1 or 2 for each of the 18 factors. Point 2 is when the shape and position of the element is accurately drawn, point 1 is when one of the shape or position is correct. Point 0.5 is when both the shape and position are incorrect, but the examinee can determine what the subject was trying to draw, and point 0 is the case when the shape and position difference are both inadequate, and when the element is not drawn. The total score is the sum of the scores scored for each of the 18 elements; It is possible scores range from 0 to 36(Higher numbers indicate better).
Change in Trail Making Test (TMT) Between Baseline and End of Treatment | Screening, baseline, day 15, day 30, day 60
  Results for both TMT A and B are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment. The reduction in the number of seconds the patients take to make the test after the study treatment means an improvement in cognitive functions.
Memory performance assessed using digit span memory test | Screening, baseline, day 15, day 30, day 60
  Digit Span Forward requires the Participant to repeat numbers in the same order as read aloud by the examiner, and Digit Span Backward requires the child to repeat the numbers in the reverse order of that presented by the examiner.
fatigue severity scale (FSS) | Screening, baseline, day 15, day 30, day 60
  The Fatigue Severity Scale (FSS) is a self-reported measure of fatigue and sleep disturbance in patients with fibromyalgia. It is a 9-item scale that assesses the severity of fatigue, the impact of fatigue on daily activities, and the degree of sleep disturbance. The FSS is a widely used instrument in research and clinical practice, and has been found to be a valid and reliable measure of fatigue and sleep disturbance in patients with fatigue and sleep disorders. The FSS items are rated on a 5-point Likert scale, with responses ranging from "not at all" to "extremely." The total score ranges from 0 to 36, with higher scores indicating greater levels of fatigue and sleep disturbance.
mental chatter 5-point scale | Screening, baseline, day 15, day 30, day 60
  Grading will be assessed on a 5-point ordinal scale. Score assessment according to the following- 1-High mental chatter, 2-Moderate mental chatter, 3-Less but frequent mental chatter, 4-less and rare mental chatter, 5-no mental chatter.
Epworth Sleepiness Scale | Screening, baseline, day 15, day 30, day 60
  How likely is the participant to doze off or fall asleep in the following situations? You should rate their chances of dozing off, not just feeling tired. Even if the participant has not done some of these things recently try to determine how it would have affected them. For each situation, decide whether or not the participant would have: · No chance of dozing =0 · Slight chance of dozing =1 · Moderate chance of dozing =2 · High chance of dozing =3 Write down the number corresponding to the choice in the right hand column.
  Interpretation: 0-7: It is unlikely that the participant is abnormally sleepy; 8-9: The participant has an average amount of daytime sleepiness; 10-15: The participant may be excessively sleepy depending on the situation. The participant may want to consider seeking medical attention; 16-24: The participant is excessively sleepy and should consider seeking medical attention.
ADHD Self-Report Scale (ASRS) | Screening, baseline, day 15, day 30, day 60
  The ASRS is an 18-item self-report screening scale used to assess adult ADHD. Each ASRS item contains a five-point scale where participants indicate how frequently they conduct themselves in the described manner; item responses can range from 'Never' to 'Very Often', where responses of 'Often' or 'Very Often' are consistent with ADHD typical dysfunction. When participant responses meet the criterion for ADHD typical dysfunction on at least 4 out of 6 screener items (denoted as 'Part A'), said participant will meet inclusion for the study. The remaining 12 ASRS items ('Part B') will be administered for use in the event that the screener criteria are met, and thus a need for further psychometric gradation arises.
COPE Questionnaire | Screening, day 60
  Problem-Focused Coping: A high score indicates coping strategies that are aimed at changing the stressful situation. High scores are indicative of psychological strength, grit, a practical approach to problem solving and is predictive of positive outcomes.
  Emotion-Focused Coping: A high score indicates coping strategies that are aiming to regulate emotions associated with the stressful situation. High or low scores are not uniformly associated with psychological health or ill health, but can be used to inform a wider formulation of the respondent's coping styles.
  Avoidant Coping: A high score indicates physical or cognitive efforts to disengage from the stressor. Low scores are typically indicative of adaptive coping.
STAI (State-Trait Anxiety Inventory) | Screening, day 60
  STAI: State-Trait-Anxiety-Inventory-Score This test consists of 20 items and assesses the current state of anxiety in relation to the current situation in which the patient is to the current situation in which the patient finds herself (State Anxiety) and the general anxiety state existing state of anxiety, which represents a part of her personality (Trait Anxiety).
  The sum score has a range from 20-80. Its interpretation with respective score are discussed below:
  mild anxiety (20 to 39); moderate anxiety (40 to 59); intense anxiety (60 to 80).
Profile of Mood State (POMS) questionnaire | Screening, day 60
  The Profile of Mood States (POMS) is a widely used instrument that measures mood using a 40 item questionnaire with each item rated using a response scale of five categories ranging from "not at all" to "Extremely". Higher score indicates worse mood. Total POMS score categories and stress inference:0-40 = A little; 81-120= Quite a lot; 41-80= Moderately; 121-160= Extremely.
Serum cortisol levels | Screening, day 15 and day 60
  The cortisol secretion will be evaluated by measuring morning serum cortisol levels.
ANTI-Vea-UGR computerized test | 0 hours, 1 hours, 4 hours and 8 hours after dosing at day 1 and day 60
  The Attentional Networks Test for Interactions and Vigilance-executive and arousal components (ANTI-Vea) is a computerized task. The task simultaneously assesses the main effects and interactions of the three attentional networks (i.e., phasic alertness, orienting, and executive control) and two dissociated components of vigilance with reasonable reliability (executive and arousal vigilance).

SECONDARY OUTCOMES:
Safety of participant assessed using adverse events. | Baseline, day 15, day 30, day 60
  It is measure in terms of No. of events.
Safety of participant Assessed using treatment compliance and tolerability of investigational product | Baseline, day 15, day 30, day 60
  It is measure in terms of percentage
Systolic blood pressure difference from reference measurement (mmHg) | Baseline, day 15, day 30, day 60
  Assessed against standard clinical grade instrument: automated oscillometric blood pressure device (mmHg
Diastolic blood pressure difference from reference measurement (mmHg) | Baseline, day 15, day 30, day 60
  Assessed against standard clinical grade instrument: automated oscillometric blood pressure device (mmHg)
Pulse rate difference from reference measurement (beats per minute) | Baseline, day 15, day 30, day 60
  Assessed against standard clinical grade instrument: Finger-based pulse oximeter (beats per minute)
Complete blood count | Screening and day 60
  White blood cell and platelet count [Thousand per microliter (Thousand/uL)] Red blood cell count [Millions per microliter (million/uL)]
Serum Glutamic Pyruvic Transaminase (SGPT) | Screening and day 60
  Blood level of SGPT was measured. (U/L)
serum glutamic-oxaloacetic transaminase (SGOT) | Screening and day 60
  Blood level of SGOT was measured. (U/L)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ramshyam Agarwal, MBBS, DNB, Principal Investigator — Lokmanya Medical Research Centre and Hospital

IPD SHARING:
Plan to Share IPD: No